CLINICAL TRIAL: NCT03390816
Title: Nutritional Status Assessment in the Elderly Suffering From Cancer (NutriAgeCancer) : a National Cross-UCOG Survey
Brief Title: Nutritional Status Assessment in the Elderly Suffering From Cancer : a National Cross-UCOG Survey
Acronym: NutriAgeCancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Société Francophone d'Onco-Gériatrie (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A01397-46
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Malnutrition; Cancer; Elderly
Keywords: malnutrition; cancer; elderly
MeSH Terms: conditions — Malnutrition; Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transversal: Elderly people, who are more than 70 years old, suffering from cancer, waiting for a treatment decision and taken care of in a hospital
  Interventions: Other: Nutritional assessment
- Longitudinal: Elderly people, who are more than 70 years old, suffering from cancer, waiting for a treatment decision and taken care of in a hospital Forward-looking follow-up of 6 months of a sub-sample during the first year
  Interventions: Other: Nutritional assessment

INTERVENTIONS:
Other: Nutritional assessment — Observational

SUMMARY:
Protein-energy malnutrition (PEM) is a frequent condition in patients suffering from cancer, especially the elderly. According to some studies, this malnutrition has important consequences in this population, by increasing the risk of treatment toxicities, premature interruption of chemotherapy, mortality and risks of complications. Identifying cases of malnutrition is an objective pursued by the National Nutrition and Health Programme and an important task of the "Unités de Coordination en Oncogériatrie".

The main goal of this study is to assess the loss of weight over the 6 month-period preceding the cancer treatment, regardless of kind (chemotherapy, targeted therapy, hormone therapy, immunotherapy, radiation therapy, surgery, comfort care), in the elderly suffering from cancer.

ELIGIBILITY:
Inclusion Criteria:

* Over 70 years of age
* Suffering from cancer
* Waiting for a treatment decision (whatever it is)
* Hospitalized in a hospital or come to consult in a hospital during the period of inclusion (2 periods of 6 weeks for two consecutive years)
* Affiliated to a social security system

Exclusion Criteria:

* Patient unable to receive information regarding the study and/or provide its non objection regarding the use of its data
* Patient under tutorship or curatorship, deprived of freedom or placed under judicial protection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly people, who are more than 70 years old, suffering from cancer, waiting for a treatment decision and taken care of in a hospital
Sampling Method: Non-Probability Sample
Enrollment: 1886 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2019-06-27 (Estimated)

PRIMARY OUTCOMES:
loss of weight | 3 to 6 month-period preceding the cancer treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elena PAILLAUD, PHD, Principal Investigator — APHP
Locations (1):
- Hôpital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No